CLINICAL TRIAL: NCT04759313
Title: Image Narrative With College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jaehee Yi, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: imagenarrative
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Depression, Anxiety
Keywords: depression; college students; posttraumatic growth; meaning making; quality of life
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imagenarrative treatment group (Experimental): INI Sessions: Each participant will take part in a 5-week program of weekly 1-hour telehealth sessions with the PI or a social work PhD student facilitator trained in the INI by the PI.
  Interventions: Behavioral: Image Narrative
- Wait List Control Group (Experimental): In weeks 6 through 10, the same program will be delivered to the wait list control group.
  Interventions: Behavioral: Image Narrative

INTERVENTIONS:
Behavioral: Image Narrative — Each participant will take part in a 5-week program of weekly 1-hour telehealth sessions with the PI or a social work PhD student facilitator trained in the INI by the PI.

SUMMARY:
The PI developed the Image Narrative Intervention (INI) based on the research using visual images in which visual images and narratives were found to support trauma survivors in narrating their experiences and in meaning making. The proposed study is the first study to test the therapeutic effect of the INI program. The investigators propose to assess, both qualitatively and quantitatively, the feasibility and preliminary effect of the INI through a pilot randomized control trial (RCT) design with a wait list control.

DETAILED DESCRIPTION:
AIM 1. To understand the unique experiences of emerging adult college students during the Covid-19 pandemic (especially around the themes of the self, relationships with others, and the future).

AIM 2. To evaluate the feasibility of the INI for emerging adult college students during the Covid-19 pandemic, both quantitatively and qualitatively.

AIM 3. To evaluate the preliminary efficacy of the INI on distress, PTG, Quality of Life and Meaning-Making.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 in age
* college students at the University of Utah
* reporting moderate or higher levels of distress in DASS21

Exclusion Criteria:

-

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
DASS (Depression, Anxiety and Stress Scale) 21 | change through study completion, an average of 3 months
  measuring distress, 0-63, higher is worse
PTGI (posttraumatic growth index) | change through study completion, an average of 3 months
  measuring posttraumatic growth, 0-105, higher is better
WHOQOL (WHO quality of life)-bref | change through study completion, an average of 3 months
  measuring quality of life, 0-100, higher is better
MLQ (meaning in life) | change through study completion, an average of 3 months
  measuring meaning making, 0-70, higher is better

CONTACTS AND LOCATIONS:
Overall Officials: Jaehee Yi, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No